CLINICAL TRIAL: NCT06691386
Title: A Randomized, Controlled, Partial-Blind, Crossover Study to Characterize the Nicotine Pharmacokinetics and Subjective Effects of Five Oral Nicotine Products Relative to Moist Smokeless Tobacco (MST) in Adult MST Users
Brief Title: Nicotine Pharmacokinetics and Subjective Effects of Oral Nicotine Products Relative to Smokeless Tobacco in Adult Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altria Client Services LLC (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: ALCS-REG-22-03-OTDN
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Tobacco Use
Keywords: Tobacco; Moist Tobacco; Oral Derived Tobacco Nicotine
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Intervention Model Description: This was a 6-way crossover design to evaluate plasma nicotine PK and subjective effects associated with the use of different nicotine levels (6, 9, and 12 mg) and different flavors of oral TDN products and subjects' OBMST product. A 6x6 Latin Square was used for the randomization, with the following sequences: Sequence 1 = ABFCED, Sequence 2 = BCADFE, Sequence 3 = CDBEAF, Sequence 4 = DECFBA, Sequence 5 = EFDACB, and Sequence 6 = FAEBDC. For pharmacokinetics analysis a linear mixed model for analysis of variance was performed on the natural log-transformed nicotine baseline-adjusted PK parameters Cmax(0-180) and AUC(0-180). For subjective effects measures a linear mixed model for analysis of variance was performed on each of the Emax-UC parameter values for the 2 items in the Smokeless Urge and Craving Questionnaire and for each of the Emax-PE parameter values for the 7 items in the Product Effects Questionnaire.
Who Masked: Participant
Masking Description: This was a partial and single-blind study. During the in-clinic product use period, subjects knew whether the product was a pouch or MST product but were blinded to the strength of the oral TDN product they used on a given day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Randomization Sequence 1 = ABFCED (Experimental): Usage of Test and Reference study products in controlled use and ad libitum use sessions during the 6 day in-clinic period in following order:
  Test Product A
  Test Product B
  Reference Product F
  Test Product C
  Test Product E
  Test Product D
  Interventions: Other: Test Product A; Other: Test Product B; Other: Test Product C; Other: Test Product D; Other: Test Product E; Other: Reference Product F: Subjects' OBMST
- Randomization Sequence 2 = BCADFE (Experimental): Usage of Test and Reference study products in controlled use and ad libitum use sessions during the 6 day in-clinic period in following order:
  Test Product B
  Test Product C
  Test Product A
  Test Product D
  Reference Product F
  Test Product E
  Interventions: Other: Test Product A; Other: Test Product B; Other: Test Product C; Other: Test Product D; Other: Test Product E; Other: Reference Product F: Subjects' OBMST
- Sequence 3 = CDBEAF (Experimental): Usage of Test and Reference study products in controlled use and ad libitum use sessions during the 6 day in-clinic period in following order:
  Test Product C
  Test Product D
  Test Product B
  Test Product E
  Test Product A
  Reference Product F
  Interventions: Other: Test Product A; Other: Test Product B; Other: Test Product C; Other: Test Product D; Other: Test Product E; Other: Reference Product F: Subjects' OBMST
- Sequence 4 = DECFBA (Experimental): Usage of Test and Reference study products in controlled use and ad libitum use sessions during the 6 day in-clinic period in following order:
  Test Product D
  Test Product E
  Test Product C
  Reference Product F
  Test Product B
  Test Product A
  Interventions: Other: Test Product A; Other: Test Product B; Other: Test Product C; Other: Test Product D; Other: Test Product E; Other: Reference Product F: Subjects' OBMST
- Sequence 5 = EFDACB (Experimental): Usage of Test and Reference study products in controlled use and ad libitum use sessions during the 6 day in-clinic period in following order:
  Test Product E
  Reference Product F
  Test Product D
  Test Product A
  Test Product C
  Test Product B
  Interventions: Other: Test Product A; Other: Test Product B; Other: Test Product C; Other: Test Product D; Other: Test Product E; Other: Reference Product F: Subjects' OBMST
- Sequence 6 = FAEBDC (Experimental): Usage of Test and Reference study products in controlled use and ad libitum use sessions during the 6 day in-clinic period in following order:
  Reference Product F
  Test Product A
  Test Product E
  Test Product B
  Test Product D
  Test Product C
  Interventions: Other: Test Product A; Other: Test Product B; Other: Test Product C; Other: Test Product D; Other: Test Product E; Other: Reference Product F: Subjects' OBMST

INTERVENTIONS:
Other: Test Product A — Use of Test Product A in controlled use and ad libitum use sessions
  Other Names: Prototype 6 mg nicotine oral TDN pouch in Wintergreen flavor
Other: Test Product B — Use of Test Product B in controlled use and ad libitum use sessions
  Other Names: Prototype 9 mg nicotine oral TDN pouch in Wintergreen flavor
Other: Test Product C — Use of Test Product C in controlled use and ad libitum use sessions
  Other Names: Prototype 12 mg nicotine oral TDN pouch in Wintergreen flavor
Other: Test Product D — Use of Test Product D in controlled use and ad libitum use sessions
  Other Names: Prototype 9 mg nicotine oral TDN pouch in Mint flavor
Other: Test Product E — Use of Test Product E in controlled use and ad libitum use sessions
  Other Names: Prototype 9 mg nicotine oral TDN pouch in Tobacco flavor
Other: Reference Product F: Subjects' OBMST — Use of Reference Product F in controlled use and ad libitum use sessions. The subjects' Own Brand Moist Smokeless Tobacco (OBMST) reference products used in this study were commercially available and had been reported by the subjects as the brands they usually consume.
  Other Names: COPENHAGEN SNUFF Fine Cut; COPENHAGEN Long Cut Mint; COPENHAGEN Long Cut; COPENHAGEN Long Cut Wintergreen; SKOAL Long Cut Mint; SKOAL Long Cut Straight; SKOAL Long Cut Wintergreen; GRIZZLY Long Cut Mint; GRIZZLY Long Cut Natural; GRIZZLY Long Cut Wintergreen

SUMMARY:
The purpose of this study was to obtain information on nicotine exposure following the use of five oral tobacco-derived nicotine (OTDN) products relative to subjects' own brand moist smokeless tobacco (OBMST) product in adult moist smokeless tobacco (MST) users, as well as to characterize subjective effects under controlled use conditions. Male and female adult MST users between the ages of 22 to 65 years were recruited. The total duration of participation for each subject was approximately 34 days including screening and a 6-day in-clinic study confinement period.

DETAILED DESCRIPTION:
This was a partial and single-blind (oral TDN products and subject only), randomized, 6-way crossover design to evaluate plasma nicotine PK and subjective effects associated with the use of different nicotine levels (6, 9, and 12 mg) and different flavors of oral TDN products (Wintergreen, Mint and Tobacco) and subjects' OBMST product. Subjects had to be regular users of one of the following OBMST products in Natural, Wintergreen, or Mint flavor variants (and a single Straight variant), and could not have rejected any of the listed flavors they did not use at the time: COPENHAGEN Fine Cut, COPENHAGEN Long Cut, SKOAL Long Cut, or GRIZZLY Long Cut.

Products used in the study were:

Product A 6 mg oral TDN pouch in Wintergreen (Test)

Product B 9 mg oral TDN pouch in Wintergreen (Test)

Product C 12 mg oral TDN pouch in Wintergreen (Test)

Product D 9 mg oral TDN pouch in Mint (Test)

Product E 9 mg oral TDN pouch in Tobacco (Test)

Product F Subject's OBMST (Reference)

Initial Screening Visit

Screening was performed within 28 days prior to Check-in (Day -1). Medical and tobacco use histories and demographic data were collected. Other screening procedures included a physical examination (including oral cavity and oropharynx), vital signs, electrocardiogram (ECG), body mass index (BMI), clinical laboratory tests (hematology, clinical chemistry, routine urinalysis), human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), and coronavirus disease 2019 (COVID-19) viral [antigen] tests, urine/saliva drug, urine/breath alcohol, cotinine screen, and serum pregnancy and follicle-stimulating hormone (FSH) tests (for females as appropriate).

Follow-up Screening and Product Trial Visit

Follow-up Screening

To ensure subjects met inclusion criteria, they took a pinch reflecting their typical quid size and used their OBMST for at least 45 minutes; cans were weighed before and after subjects selected their pinch size. Subjects were allowed to "top off" their pinch within the first minute, after which the total mass used was recorded; the brand of MST product used was collected. Tobacco cessation information was provided. Subjects who responded negatively (i.e., unwilling to use and/or could not tolerate their OBMST for at least 45 minutes) did not continue in the study.

Product Trial:

Following completion of screening procedures, eligible subjects participated in a product trial at home for at least 5 days and were provided a single 14-pouch can of each of the five oral TDN products to be used ad libitum prior to Day -1 to allow subjects to become accustomed to the products. Subjects who responded negatively (i.e., unwilling to use and/or could not tolerate any of the oral TDN products [e.g., experience AEs during the use of the oral TDN product that prevented them from continuing to use the product as judged by the Investigator]) to any of the study products during the Product Trial did not continue in the study.

Check-in and Randomization

Subjects who met all inclusion criteria and none of the exclusion criteria checked in to the clinic on Day -1 at a time determined by the clinic. Subjects received a COVID-19 viral [antigen] test. Female subjects received a pregnancy test as well. Subjects demonstrated that they were able/willing to use the 12 mg nicotine product (Product C) by using one pouch for at least 45 minutes. The 12 mg demonstrated use session had to be completed at least 4 hours prior to the start of the first ad libitum use session. Subjects were trained on the questionnaires for familiarization with the questions, scales, and computerized tablets prior to randomization by completing the questionnaires during a training session.

Subjects were randomized to 1 of 6 product sequences on Day -1 prior to the afternoon ad libitum product use episode. A 6x6 Latin Square was used for randomization, with the following sequences: Sequence 1 = ABFCED, Sequence 2 = BCADFE, Sequence 3 = CDBEAF, Sequence 4 = DECFBA, Sequence 5 = EFDACB, and Sequence 6 = FAEBDC. Subjects were stratified based on age (Males only [Low (<45), High (≥46)]) and sex.

A total of 64 subjects (63 males, 1 female) were enrolled and 56 subjects (55 males, 1 female) were ultimately randomized to one of six study product sequences. Subjects were not allowed to use any tobacco/nicotine-containing product other than the assigned ones from the time of Check-in on Day -1 through the completion of last study procedure on Day 6.

Ad Libitum Product Use (Afternoon Use Session)

On each of Days -1 through 5, subjects participated each afternoon, starting at least 2 hours after the last PK blood draw, as applicable, but no later than 16 hours prior to the following morning's controlled product use, in an approximately 2-hour (± 10 minutes) ad libitum product use episode. Subjects were allowed to use up to 2 units (oral TDN pouch or OBMST quid) of the same product as the assigned product for the following morning's controlled product use episode per randomization.

Controlled Product Use (Pharmacokinetic Use Session)

On the morning of each study day (Days 1 - 6), subjects used the assigned product under controlled conditions:

* Oral TDN product (Products A, B, C, D, and E): use one unit of oral TDN product by placing the product in the mouth at the location chosen by the subject for 45 minutes.
* OBMST product (Product F): use one quid of the OBMST by placing the product in the mouth at the location chosen by the subject for 45 minutes. The quid mass for each subject was determined at Screening, and was weighed to ± 0.1 g.

Used oral TDN products and expectorate from the OTDN controlled product use episodes were collected; the used MST quids were discarded.

PK Blood Sample Collection

On Days 1 through 6, venous blood samples (~4 mL) for nicotine PK were collected at 5 minutes prior to, and at 5, 15, 30, 40, 45, 50, 60, 90, 120, and 180 minutes following the start of each controlled product use episode. Used study products were collected (with the exception of the OBMST) for analysis of residual nicotine.

Subjective Effects Measures

For collection of primary outcome measures subjects completed the following subjective measures questionnaires:

* Smokeless Urge and Craving Questionnaire before, during, and following each controlled product use episode
* Product Effects Questionnaire during and following each controlled product use episode

Available data from all 56 randomized subjects (55 males, 1 female) were included in the analysis of primary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary consent to participate in this study documented on the signed informed consent form (ICF).
* Adult males and females 22 to 65 years of age, inclusive, at Screening. Full COVID-19 vaccination (FDA authorized vaccines) record that was completed at least 14 days prior to Screening for subjects >45 years of age. Full vaccination as defined by the Centers for Disease Control and Prevention.
* Self-affirmed adult consumers of MST with usual brand of COPENHAGEN Fine Cut, or COPENHAGEN Long Cut, SKOAL Long Cut, or GRIZZLY Long Cut MST products in Mint, Natural, and Wintergreen flavor variants (and a single Straight variant; consumption of at least ½ can per day in the 30 days prior to Screening) for at least 12 months prior to Check-in; subjects cannot reject any of the flavor variants. Brief periods (i.e., up to 7 consecutive days) of non-MST usage within 90 days before Check-in (e.g., due to illness, participation in a clinical study where tobacco use was prohibited) will not be exclusionary at the discretion of the Investigator.
* Positive urine cotinine (≥ 500 ng/mL) at Screening.
* Negative pregnancy test at Screening, prior to the start of Product Trial, and Check-in (Day -1) for all female subjects.
* Female subjects who are heterosexually active and of childbearing potential (e.g., not surgically sterile at least 6 months prior to Check-in nor postmenopausal with amenorrhea for at least 1 year prior to Check-in and FSH levels consistent with postmenopausal status) must have been using one of the following forms of contraception and agree to continue using it through completion of the study:

  * hormonal (e.g., oral, vaginal ring, transdermal patch, implant, injection) consistently for at least 3 months prior to Check-in,
  * double barrier (e.g., condom with spermicide or diaphragm with spermicide) consistently for at least 2 weeks prior to Check-in,
  * intrauterine device for at least 3 months prior to Check-in,
  * exclusive partner who has been vasectomized for at least 6 months (inclusive) prior to Check-in.

Female subjects of childbearing potential who are not currently engaging in heterosexual intercourse must agree to use one of the above methods of birth control through completion of study, in the event that they have heterosexual intercourse during the course of the study.

* Female subjects who are of nonchildbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to Check-in:

  * hysteroscopic sterilization with documentation of success with hysterosalpingogram;
  * bilateral tubal ligation or bilateral salpingectomy;
  * hysterectomy;
  * bilateral oophorectomy; or be postmenopausal with amenorrhea for at least 1 year prior to Check-in and have FSH levels consistent with postmenopausal status.
* Willing to comply with the requirements of the study.
* Willing and able to use all oral TDN study products for at least 45 minutes.

Exclusion Criteria:

Subjects will be excluded from the study if there is evidence of any of the following criteria at Screening or Check-in, or at any time during the study as appropriate.

* An ad libitum pinch mass that is less than 2 g as captured at the Follow-up Screening visit.
* Use of any oral TDN or nicotine-containing products with the exception of MST and combustible cigarettes (e.g., nicotine lozenge, nicotine gum, nicotine inhaler, nicotine mouth spray, nicotine pouch) within the past 30 days prior to the screening visit.
* Any postponement of a quit attempt in order to participate in the study.
* Attempts to quit MST product use in the 3 months prior to Day -1 (Check- in).
* Planning to quit MST product use in the next 3 months (from Screening visit).
* Negative response (i.e., unwilling to use or unable to tolerate [e.g., experiences AEs during the Product Trial that will prevent them from continuing to use the product as judged by the Investigator]) to any of the oral TDN study products during the Product Trial.
* Dentition that prevents subjects from using products.
* History or presence of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, urologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
* Clinically significant abnormal findings on the vital signs, physical examination (including oral cavity and oropharynx), medical history, or clinical laboratory results, in the opinion of the Investigator.
* Positive test for HIV, HBsAg, COVID-19 or HCV at Screening or Check-in, as applicable.
* History or presence of any type of malignant tumors.
* Current evidence or any history of congestive heart failure.
* Diabetes mellitus that is not controlled by diet/exercise alone, in the opinion of the Investigator. Fasting serum glucose of 126 mg/dL [7 mmol/L] is exclusionary. One re-check may be performed for values greater than or equal to 126 mg/dL but less than 200 mg/dL.
* An acute illness (e.g., upper respiratory infection, viral infection) requiring treatment with prescribed medicines within 2 weeks prior to Check-in or at the discretion of the Investigator.
* Presence of gum bleeding and/or abscess, open mouth sores or oral ulcers at Screening or Check-in.
* Allergic to or cannot tolerate mint, cool mint, spearmint, or peppermint flavoring agents.
* Any planned surgery from the time of Screening through the End-of-Study.
* History of drug or alcohol abuse within 24 months prior to Check-in.
* Fever (i.e., body temperature > 100.5 ͦ F) at Screening or Check-in. One re-check may be performed at the Investigator's discretion.
* Systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 90 mmHg at Screening or Check-in, measured after being seated for at least 10 minutes. Two re-checks may be performed at the Investigator's discretion.
* BMI greater than 40.0 kg/m2 or less than 18.0 kg/m2 at Screening.
* Estimated glomerular filtration rate (eGFR) < 80 mL/minute (using the Modification of Diet in Renal Disease formula) at Screening.
* Serum alanine aminotransferase (ALT) ≥ 1.5 times the upper limit of normal and/or aspartate aminotransferase (AST) ≥ 2.0 times the upper limit of normal at Screening.
* Positive urine/breath screen for alcohol at Screening or Check-in.
* Positive urine/saliva screen for any of the following drugs of abuse, regardless of the reason of use: amphetamines, opiates, cannabinoids, or cocaine at Screening or Check-in.
* Female subjects who are pregnant (positive serum/urine pregnancy test at Screening, prior to the start of Follow-up Screening/Product Trial, or Check-in), lactating, or intend to become pregnant from Screening through the End-of-Study.
* Use of medications known or are suspected to interact with cytochrome P450 2A6 (including, but not limited to, amiodarone, amlodipine, amobarbital, buprenorphine, clofibrate, clotrimazole, desipramine, disulfiram, entacapone, fenofibrate, isoniazid, ketoconazole, letrozole, methimazole, methoxsalen, metyrapone, miconazole, modafinil, orphenadrine, pentobarbital, phenobarbital, pilocarpine, primidone, propoxyphene, quinidine, rifampicin, rifampin, secobarbital, selegiline, sulconazole, tioconazole, tranylcypromine) within 14 days or 5 half-lives of the drug, whichever is longer, prior to Check-in or during the study.
* Use of antibiotic treatment within 2 weeks prior to Check-in.
* Plasma donation within 7 days prior to Day 1.
* Donation of blood or blood products (with the exception of plasma as noted above), had significant blood loss, or received whole blood or a blood product transfusion within 56 days prior to Day 1.
* Participation in a previous clinical study for an investigational drug, device, biologic, or for a tobacco product within 30 days prior to Check- in.
* Participation in more than two Altria Client Services LLC (ALCS) sponsored studies within the past 12-month period prior to Check-in.
* Subject or a first-degree relative (i.e., parent, sibling, child, spouse) is a current or former employee of the tobacco industry or a named party or class representative in litigation with any tobacco company.
* Subject or a first-degree relative (i.e., parent, sibling, child, spouse) is a current employee of the study site.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Plasma Nicotine (ng/mL) | Day 1 through Day 6
  Maximum plasma nicotine concentration (Cmax) measured following the product use under controlled use conditions
Smokeless Urge and Craving Questionnaire | Day 1 through Day 6
  Maximum reduction in response relative to pre-use for subjective ratings of all items in the Smokeless Urge and Craving Questionnaire (Emax-UC) following the product use under controlled use conditions. Each question was paired with a 100 millimeter (mm) visual analog scale (VAS). The VAS was anchored with "Not at All" on the left and "Extremely on the right. Subjects placed a vertical line at a place along the VAS based on how he/she felt in the moment. Scoring of response based on measurement of distance in mm from "Not at All" hash to mark made by subject with no response being better or worse.
Product Effects Questionnaire | Day 1 through Day 6
  Maximum response for subjective ratings of all items in the Product Effects Questionnaire (Emax-PE) following the product use under controlled use conditions. Each question was paired with a 100 millimeter (mm) visual analog scale (VAS). The VAS was anchored with "Not at All" on the left and "Extremely" on the right. Subjects placed a vertical line at a place along the VAS based on how he/she felt in the moment. Scoring of response based on measurement of distance in mm from "Not at All" hash to mark made by subject with no response being better or worse.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Pillar Clinical Research LLC, Bentonville, Arkansas
  - QPS Bio-Kinetic, Springfield, Missouri

IPD SHARING:
Plan to Share IPD: No